CLINICAL TRIAL: NCT05281367
Title: The Effect of Facilitated Tucking, Maternal Breast Milk Odor and Non Nutritive Sucking During Heel Stick on Procedural Pain in Premature Neonates
Brief Title: Non-pharmacological Methods in Pain Managment During Heel Stick in Preterm Infants
Acronym: (pain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Negarin Akbari (Other)
Responsible Party: Sponsor-Investigator, Negarin Akbari, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1400829255739
Record Dates: First submitted 2022-01-18; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pain, Acute; Neonatal Intensive Care Unit
MeSH Terms: conditions — Acute Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breast milk odor group (Experimental): It is a non-pharmacological method of pain control in which 3 cc of breast milk will be dripped onto a sterile pad and It will be placed at a distance of 10 cm from the nose of the newborn. Precisely, premature newborns' own mothers' milk will be used. For this, mothers of newborns will be contacted and breast milk will be provided for the day of the procedure.
  Interventions: Procedure: Breast milk odor group
- Facilitated tucking group (Experimental): It is a non-pharmacological method of pain control in which the arms and legs are slowly contracted and placed close to the body. In this method, the baby is placed on its side, the baby's back is gently bent, the legs are folded at an angle of more than 90 degrees, the shoulders are folded up to 90 degrees, and the care hands are placed either on the head near the mouth or Placed on the baby's face.
  Interventions: Procedure: Facilitated tucking group
- Non-nutritive sucking group (Experimental): It is a non-pharmacological method used to control pain in infants. In this method, babies suck without receiving the nutrient. This can be done by a pacifier, a parent's hand or a nurse.
  Interventions: Procedure: Non-nutritive sucking group
- control grup (Experimental): The control group will consist of 36 premature newborns who are routinely applied in the clinic. In the clinic where the research was conducted, no attempt is made to reduce pain during heel stick.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Breast milk odor group — The researcher applied the breast milk that dripped on the pad for 3 minutes before the heel stick for 36 premature newborns in the breast milk odor group. About three cc breast milk dripped onto a sterile pad and placed at a distance of 10 cm from the nose of the newborn. It continued until 3 minutes after the invasive procedure. Heart rate, arterial oxygen saturation, and respiration rate were recorded in this group before the study. Then, to evaluate the pain in the infants, a video camera was placed on the incubator. The infants in each group were filmed from three minutes before the procedure to three minutes after. Neonatal pain was measured at 1, 2, and 3 minutes before, during, and at 1, 2, and 3 minutes after the procedure by two researchers independently using the new version Premature Infant Pain Profile (PIPP).
  Other Names: Breast milk odor
  Arms: Breast milk odor group
Procedure: Facilitated tucking group — The Facilitated tucking position was given to 36 premature newborns in the Facilitated tucking group, from 3 minutes before to 3 minutes after the heel stick procedure. Premature newborns were kept in the facilitated tucking position by the investigator using the incubator windows without opening the incubator cover to prevent heat loss of the newborn. Heart rate, arterial oxygen saturation, and respiration rate were recorded in this group before the study. Then, to evaluate the pain in the infants, a video camera was placed on the incubator. The infants in each group were filmed from three minutes before the procedure to three minutes after. Neonatal pain was measured at 1, 2, and 3 minutes before, during, and at 1, 2, and 3 minutes after the procedure by two researchers independently using the new version Premature Infant Pain Profile (PIPP).
  Arms: Facilitated tucking group
Procedure: Non-nutritive sucking group — 36 premature newborns who were in the non-nutritive sucking group were given a silicone pacifier suitable for the week of the baby's mouth from 3 minutes before to 3 minutes after the heel stick. Heart rate, arterial oxygen saturation, and respiration rate were recorded in this group before the study. Then, to evaluate the pain in the infants, a video camera was placed on the incubator. The infants in each group were filmed from three minutes before the procedure to three minutes after. Neonatal pain was measured at 1, 2, and 3 minutes before, during, and at 1, 2, and 3 minutes after the procedure by two researchers independently using the new version Premature Infant Pain Profile (PIPP).
  Other Names: pacifire
  Arms: Non-nutritive sucking group
Procedure: Control group — The control group will consist of 36 premature newborns who are routinely applied in the clinic. In the clinic where the research was conducted, no attempt is made to reduce pain during heel stick. Heart rate, arterial oxygen saturation, and respiration rate were recorded in this group before the study.
  Then, to evaluate the pain in the infants, a video camera was placed on the incubator. The infants in each group were filmed from three minutes before the procedure to three minutes after. Neonatal pain was measured at 1, 2, and 3 minutes before, during, and at 1, 2, and 3 minutes after the procedure by two researchers independently using the new version Premature Infant Pain Profile (PIPP).
  Arms: control grup

SUMMARY:
Aims and objectives: This study was performed to examine the effects of Non-nutritive sucking, breast milk odor, and Facilitated tucking on preterm infant pain before, during, and after heel-stick procedures.

Design: A randomized clinical trial in a single center.

Methods:

The study was conducted on 144 premature infants with a gestational age of 31 to 36 weeks and 6 days hospitalized in the neonatal intensive care unit of Shahid Sayad Shirazi Hospital in Iran. Neonates were randomly assigned to four groups: 36 babies were included in the Non-nutritive sucking(1st Group), 36 in breast milk odor (2nd Group), 36 in Facilitated tucking (3rd Group), and 36 in the control group (4th Group). Pain score, heart rate, oxygen saturation, and respiratory rate of the babies in all groups before, during, and after the procedure were evaluated by two nurses independently.

DETAILED DESCRIPTION:
Aim: Due to the necessity of various painful procedures and their side effects on infants, pharmacological and non-pharmacological methods are adopted to reduce the pain. Since pharmacological methods can be associated with several side effects, it is better to use non-pharmacological methods for pain control in newborns. Therefore, the purposes of this study were to compare the effects of three different methods (including Non-nutritive sucking, breast milk odor, and Facilitated tucking) on preterm infant pain before, during, and after heel-stick procedures.

Method: The study was conducted on 144 premature infants with a gestational age of 31 to 36 weeks and 6 days hospitalized in the neonatal intensive care unit of Shahid Sayad Shirazi Hospital, Iran. Initially, neonates are divided into two groups according to gestational age (including neonates between 31-33 weeks and 34-36 weeks) to moderate the confounding effect of the age, and then the allocation of neonates to four groups was performed.

Using the stratification block randomization method, 36 babies were included in the Non-nutritive sucking(1st Group), 36 in breast milk odor (2nd Group), 36 in Facilitated tucking (3rd Group), and 36 in the control group (4th Group). Two researchers viewed the recorded videos independently and evaluate the heart rate, oxygen saturation, respiratory rate, and neonatal pain at 1st,2nd,3rd minute before the procedure, during, and at 1st,2nd,3rd minutes after the procedure according to the Premature Infant Pain Profile (PIPP).

ELIGIBILITY:
Inclusion Criteria:

1. Week of gestation is between 31 and 36 weeks
2. Not being exposed to a painful procedure at least 1 hour before the interventions
3. At least 1 hour has passed since feeding
4. Not taking analgesics and/or sedatives in the last 4 hours
5. Body weight of 1000 grams or more
6. Having mother's milk
7. Not exceeding the 10th day of postnatal age

Exclusion Criteria:

1. Having ventilator support
2. Having a congenital anomaly
3. Using analgesic / narcotic analgesic drugs
4. Continuous sedative treatment
5. Having a congenital malformation that may cause asphyxia and affect respiration
6. Having intracranial bleeding

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 1 minutes before the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 2 minutes before the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 3 minutes before the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured during the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 1 minutes after the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 2 minutes after the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.
Pain score of preterm infants assessed on the Premature Infant Pain Profile Revised (PIPP-R) | Pain was measured at 3 minutes after the procedure by two researchers independently.
  PIPP is a valid instrument that can be used to assess infants' response to pain. The instrument estimates the baby's pain based on assigning a score of zero to four to each of the fetal ages, behavioral status, maximum heart rate, minimum oxygen saturation, eyebrow bulges, eye presses, lip and nose creases. This tool's minimum and maximum pain scores are zero and 21, respectively.

SECONDARY OUTCOMES:
Heart rate during heel stick | from 4 minutes before heel stick to 4 minute after heel stick
  Heart rate initially was recorded in each group 4 minutes before starting any intervention. Then, 1,2, and 3 minutes before heel stick, During heel stick, and 1,2,3 minutes after heel stick it again measured (totally eight times).
Respiratory rate | From 4 minutes before heel stick to 4 minute after heel stick
  Respiratory rate initially was recorded in each group 4 minutes before starting any intervention. Then, 1,2, and 3 minutes before heel stick, During heel stick, and 1,2,3 minutes after heel stick it again measured (totally eight times).
Oxygen saturation | From 4 minutes before heel stick to 4 minute after heel stick
  Oxygen saturation initially was recorded in each group 4 minutes before starting any intervention. Then, 1,2, and 3 minutes before heel stick, During heel stick, and 1,2,3 minutes after heel stick it again measured (totally eight times).

OTHER OUTCOMES:
Crying time | During procedure (During heel stick the total crying time was measured from where it starts until the over.)
  The researcher recorded the crying time in second (sec) during heel stick.

CONTACTS AND LOCATIONS:
Overall Officials: Negarin Akbari, PhD student, Principal Investigator — Istanbul un'vers'ty cerrahpasa-Istanbul,Turkey
Locations (1):
- Golestan University of Medical Sciences, Gorgan, Golestan Province, Iran

IPD SHARING:
Plan to Share IPD: No